CLINICAL TRIAL: NCT02631759
Title: Prevention of Epileptic Seizures in Acute intraCerebral Haemorrhage
Acronym: PEACH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014-845
Record Dates: First submitted 2015-12-07; First posted 2015-12-16 (Estimated); Last update posted 2025-09-26 (Actual); Status verified 2022-04

CONDITIONS: Acute intraCerebral Haemorrhage
Keywords: Acute intraCerebral Haemorrhage, Epileptic seizures, Lévétiracetam
MeSH Terms: conditions — Seizures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lévétiracetam (Experimental): 52 patients will be recruited over 2 years in the experimental group
  Interventions: Drug: Lévétiracetam
- Placebo (Placebo Comparator): 52 patients will be recruited over 2 years in the control group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lévétiracetam — Levetiracetam will be administered at 500mg / 12h through IV started within 24 hours after enrollment in the study for at least 48 hours and for up to 5 days, then a per os administration will be made out as soon as oral will be possible, at a dose of 500mg / 12h (1g / day in two divided doses ) .
  The total duration of treatment will be 1 month and 15 days taking into account the processing taking decay phase.
  The decay phase takes place in two phases:
  * A phase of 7 days of levetiracetam 250 mg every 12 hours ( morning and evening)
  * Then a phase of 7 days of levetiracetam 250 mg every 24 hours (evening).
  Arms: Lévétiracetam
Drug: Placebo — Placebo (NaCl 0,9%) will be administered at 500mg / 12h through IV started within 24 hours after enrollment in the study for at least 48 hours and for up to 5 days, then a per os administration will be made out as soon as oral will be possible, at a dose of 500mg / 12h (1g / day in two divided doses ) .
  The total duration of treatment will be 1 month and 15 days taking into account the processing taking decay phase.
  The decay phase takes place in two phases:
  * A phase of 7 days of placebo 250 mg every 12 hours ( morning and evening)
  * Then a phase of 7 days of placebo 250 mg every 24 hours (evening).
  Arms: Placebo

SUMMARY:
Haemorrhagic strokes represent about 10-15 % of all strokes and 30,000 cases per year in France. The 30-day death rate ranges from 30 to 55% (50% of deaths occurring within 48 hours). Currently, no urgent medical or surgical treatment has been shown to improve functional or vital prognosis. Clinical epileptic seizures frequency in acute intracerebral haemorrhage has been estimated between 4% and 16% but the occurrence of subclinical epileptic seizures (detected on the electroencephalogram (EEG) only) could be much more frequent (28 % to 40 %).

Some studies have suggested that early repeated epileptic seizures may be associated with a worse neurological prognosis. Repeated epileptic seizures occurring in the acute phase may increase brain oedema, worsen, hypoxia and may lead to cellular death in the injured brain tissue. Thus, prevention of early epileptic seizures may improve neurological outcome. However, the efficacy of a systematic prophylactic antiepileptic treatment on clinical and subclinical epileptic seizures has not been evaluated in the setting of intracerebral haemorrhage. The current European guidelines recommend the use of antiepileptic drugs only when epileptic seizures occur.

Primary objective: PEACH is a randomized controlled trial aiming at evaluating the impact of systematic prophylactic antiepileptic treatment with levetiracetam versus placebo in acute supratentorial spontaneous intracerebral haemorrhage. The primary endpoint is the occurrence of at least one clinical or electrical epileptic seizure recorded on continuous 48h holter EEG.

Secondary Objectives:This study also aims to assess:

Ä The efficacy of prophylactic treatment with levetiracetam on the number of EEG seizures, on the total duration of epileptic seizures continuously recorded on EEG, on the occurrence of some paroxysmal EEG patterns, on the number of clinical seizures occurred during 72 hours of diagnosis, on the occurrence of early (day-0 to day-30 ) and late (from day-30 to 12 months) clinical seizures, on the functional prognosis at 3 , 6 and 12 months evaluated by the modified Rankin scale , on the cerebral oedema and mass effect evaluated by comparing the admission brain CT scan with the control CT scan performed at 72 hours, on the neurological status as assessed by the National Institute of Health Stroke Scale at 72 hours , 1 month and 3 months and on the quality of life measured by the Stroke impact Scale at 3, 6 and 12 months.

Ä The frequency of side effects related to treatment with levetiracetam (anxiety and depression assessed by the Hospital Anxiety and Depression Scale at 1 and 3 months) Sample Size: 104 patients will be recruited over 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years with no upper age limit
* Competent adult patient.
* Patient affiliated to the French National Health Insurance.
* Patient with supratentorial spontaneous intracerebral hemorrhage diagnosed by CT or MRI
* Early neurological symptoms less than 24 hours
* NIHSS score on admission between 5 and 25
* Informed consent given by the patient or his legal representative

Exclusion Criteria:

* Inaugural Seizures ( at the onset of symptoms associated with intracerebral hemorrhage )
* Seizures occurring between the inclusion of the patient and the start of the EEG
* Other Intracerebral hemorrhage infratentorial , post-traumatic , related to a vascular malformation or an underlying tumor and secondarily hemorrhagic cerebral infarction
* Current antiepileptic treatment when intracerebral hemorrhage , or a history of epilepsy
* Modified Rankin Scale before intracerebral hemorrhage > 1 (indicating a preexisting disability)
* Serious illness which can affect the prognosis within 3 months
* Severe renal impairment ( creatinine clearance <30 ml / min)
* Pregnancy, lactation
* Known hypersensitivity to levetiracetam or other pyrrolidone derivatives , or any of the excipients.
* Untreated severe depression , psychotic disorders
* Lactose Intolerance
* Patient under measuring socio- legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2021-06-07 (Actual)

PRIMARY OUTCOMES:
Occurrence of at least one clinical or electrical epileptic seizure recorded on continuous 48 hours holter EEG | 48 hours

SECONDARY OUTCOMES:
Occurrence of electroencephalographic signs | 48 hours
Number of EEG seizures | 48 hours
Total duration of epileptic seizures continuously recorded on EEG | 48 hours
occurrence of some paroxysmal EEG patterns | 48 hours

OTHER OUTCOMES:
Occurrence of early (day-0 to day-30 ) and late (from day-30 to 12 months) clinical seizures | 12 months
Functional prognosis at 3 , 6 and 12 months evaluated by the modified Rankin scale | 12 months
Cerebral oedema and mass effect evaluated by comparing the admission brain CT scan with the control CT scan performed at 72 hours | 72 hours
Neurological status as assessed by the National Institute of Health Stroke Scale at 72 hours , 1 month and 3 months | 3 months
Quality of life measured by the Stroke impact Scale at 3, 6 and 12 months | 12 months
frequency of side effects related to treatment with levetiracetam (anxiety and depression assessed by the Hospital Anxiety and Depression Scale at 1 and 3 months) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Laure Peter-Derex, MD, Study Director — Hospices Civils de Lyon
Locations (1):
- Department of functional neurology and epileptology, Lyon, France

REFERENCES:
- [Result] Peter-Derex L, Philippeau F, Garnier P, Andre-Obadia N, Boulogne S, Catenoix H, Convers P, Mazzola L, Gouttard M, Esteban M, Fontaine J, Mechtouff L, Ong E, Cho TH, Nighoghossian N, Perreton N, Termoz A, Haesebaert J, Schott AM, Rabilloud M, Pivot C, Dhelens C, Filip A, Berthezene Y, Rheims S, Boutitie F, Derex L. Safety and efficacy of prophylactic levetiracetam for prevention of epileptic seizures in the acute phase of intracerebral haemorrhage (PEACH): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Neurol. 2022 Sep;21(9):781-791. doi: 10.1016/S1474-4422(22)00235-6. PMID 35963261